CLINICAL TRIAL: NCT04363112
Title: Association Between a Biological Pattern of Dysregulation of the HPA Axis and Mental Disorders in Children Exposed to Early Life Stress
Acronym: ESASP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitement difficulties
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 29BRC20.0056
Record Dates: First submitted 2020-04-20; First posted 2020-04-27 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-07

CONDITIONS: Mental Disorder, Child
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: The study is an monocentric, interventional, comparative uncontrolled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study with just one arm (Other): All of participants are in this arm. Mini Kid II and CBCL score are administered between day 3 and 7. Moreover, salivary test will be remove to evaluate cortisol secretion, 4 time per day during 2 consecutive days.
  Psychologic aftercare will be propose if children have psychologic troubles (results of Mini Kid II)
  Interventions: Behavioral: Mini Kid II

INTERVENTIONS:
Behavioral: Mini Kid II — Mini Kid II (Mini International Neuropsychiatric Interview ) is a standardised, hetero mental health questionary for children, according to DSM IV. Mini Kid II will be administered to children between day 3 and 7 during the study.

SUMMARY:
The purpose of this study is to demonstrate an association between a biological pattern of dysregulation of the HPA axis and mental disorders in children exposed to early life stress.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate an association between a biological pattern of dysregulation of the HPA axis and mental disorders in children exposed to early life stress.

Cortisol secretion lead to define two groups : pathologic versus normal cortisol secretion.

Mental disorders is evaluate with Mini-Kids II (a mental health questionary) and lead to define two groups : mental disorders versus no mental disorders

ELIGIBILITY:
Inclusion Criteria:

* Aged 8 to over 10 years
* To be entrust to ASE of Finistère in stable environment (the same place of residence since 6 months or more)
* French speaking
* Oral consent by children
* Informed and signed consent by tenured of parent authority

Exclusion Criteria:

* Don't want to participate
* To have chronic neurologic or endocrinal pathology or don't have access to verbal language.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Mini Kid II : Mini International Neuropsychiatric Interview | Day 10 to the study
  Standardized questionary administered by a physician. There are 30 pages with 17 subjects like depression, maniac trouble, panic trouble, etc.

SECONDARY OUTCOMES:
CBCL score : Child Behaviour Check List | Day 10 to the study
  CBCL Score is a hetero scale administered by host family or caseworker. It is a scale 0 (no behavior troubles) to 124 (behavior troubles).
BRIEF : Behavrioral Rating Inventory of Executive Function | Day 10 to the study
  Standardized questionary administered by by host family or caseworker between day 4 and 13 to the study. BRIEF questionary contains 2 themes (metacognition and Behavior regulation) with 85 items in total. Each item contains 3 answers : Never (0)/ Sometime(1)/ Always(2)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest University Hospital. Requestors will be required to sign and complete a data access agreement.